CLINICAL TRIAL: NCT03371550
Title: Cisplatin-Docetaxel Induction Plus Concurrent 3-D Conformal Radiotherapy and Weekly Chemotherapy for Locally Advanced Non-Small Cell Lung Cancer Patients: A Phase II Trial
Brief Title: A Phase II Trial of Cisplatin-Docetaxel Induction Plus Concurrent 3-D Conformal Radiotherapy and Weekly Chemotherapy
Acronym: TAXCIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/07
Record Dates: First submitted 2017-11-30; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Locally Advanced Non-small Cell Lung Cancer
Keywords: Concurrent 3-D chemoradiotherapy,Docetaxel,Cisplatin,Chemotherapy ·
MeSH Terms: interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Intervention Model Description: This was a prospective, open-label, multicentric, phase II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiochemotherapy (Experimental): Induction chemotherapy with docetaxel and cisplatine and concomitant radiotherapy
  Interventions: Drug: Docetaxel; Radiation: concomitant radiotherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Docetaxel — Induction chemotherapy
Radiation: concomitant radiotherapy — Pulmonary and mediastinal radiotherapy
Drug: Cisplatin — Induction chemotherapy

SUMMARY:
Concurrent chemoradiotherapy (CHRT) is the standard of care for unresectable locally advanced stage III non-small cell lung cancer. However, the optimal combination remains unclear. The aim of this study is to evaluate the efficacy of 2 induction chemotherapy cycles (days 1 and 22) with docetaxel 75 mg/m2 and cisplatin 75 mg/m2 followed by concurrent chemotherapy (weekly docetaxel-cisplatin, 20 mg/m2) and 3-D conformal radiotherapy for 6 weeks (66 Gy/5 fractions per week/2 Gy per fraction). ). The primary endpoint is the response rate. Secondary objectives are toxicity, time to progression, and overall survival.

DETAILED DESCRIPTION:
Lung cancer is the most common malignancy among men in most countries and constitutes the leading cause of cancer death worldwide. Non-small cell histology represents roughly 80% of lung cancer cases comprising one third of patients with stage III, locally-advanced disease at diagnosis. Some stage IIIA cancers are considered resectable but many stage IIIA (with bulky N2) and stage IIIB (T4 any N M0, any T N3M0) cancers are considered unsuitable for surgery. However, some authors have shown that surgery after chemoradiotherapy (CHRT) is beneficial for at least progression-free survival (PFS). Since the 90s, CHRT has become the cornerstone of inoperable locally advanced non-small cell lung cancer (NSCLC). A meta-analysis of 52 randomized studies showed a survival improvement of 3% at 2 years and 2% at 5 years for patients treated with CHRT versus radiotherapy alone [6]. Concomitant chemoradiation was demonstrated to be better than sequential administration in terms of overall survival (OS) in 3 out of 4 randomized studies with esophagitis as the dose-limiting toxicity. Nevertheless, the median survival was around 16 months and improvement is needed. To better control micrometastatic disease and reduce distant relapses, one possibility is to increase radiosensitization with higher doses of chemotherapy.The aim of this phase II study is to evaluate the anti-tumoral activity of a weekly docetaxel-cisplatin combination administered concurrently with radiotherapy after 2 induction cycles with the same drugs.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed NSCLC,
* stage IIIB (excluding malignant pleural or pericardial effusions, tumoral volume exceeding one radiation field,
* N3 supraclavicular, and contralateral hilar nodal involvement) or inoperable stage IIIA defined by the new International Staging System [21],
* 18 ≤ age ≤ 75 years,
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤2,
* weight loss <10%,
* at least one measurable lesion according to RECIST 1.0 criteria,
* adequate hematopoietic function (absolute neutrophil count ≥2 × 109/l, platelets ≥100 × 109/l, and hemoglobin level ≥10g/dl), adequate hepatic function [total serum bilirubin less than or equal to the institutional upper limit of normal (ULN), aspartate aminotransferase ≤1.5× ULN, and alkaline phosphatase ≤5× ULN], and adequate renal function (serum creatinine ≤1.5× ULN).

Exclusion Criteria:

* patients previously treated with radiotherapy or chemotherapy for NSCLC,
* previous cancer except basocellular carcinoma and in situ carcinoma of the cervix curatively treated and other cancers curatively treated for at least 5 years,
* peripheral neuropathy NCI-CTC grade ≥2,
* noncontroled severe disease,
* pregnant or breast-feeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-08-05 (Actual); Primary Completion 2010-10-31 (Actual); Study Completion 2011-10-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the antitumor activity of Docetaxel - Cisplatin and concomitant thoracic radiotherapy after Docetaxel - Cisplatin induction chemotherapy in patients with locally advanced non-operable NSCLC by tumor response rate | up to 3 years
  Tumor Response rate between 6 and 8 weeks according to RECIST 1.0 criteria after the end of radiotherapy (except in the case of early progression) that patients:
  * having received at least 4 weekly injections of Docetaxel and Cisplatin,
  * who have received the full radiotherapy treatment (except in case of cessation for toxicity, in which case the patients will be evaluable).

SECONDARY OUTCOMES:
Overall survival and at 12 months | up to 3 years
  To evaluate the overall survival at 12 months between the first day of treatment to the death
Response delay | up to 3 years
  Complete response delay evaluated between the day of the complete response to the progression and partial response between the first day of the treatment and the progression
Progression Free Survival | up to 3 years
  To evaluate Progression free survival according to RECIST criteria
Tolerance profile of the association in terms of immediate and delayed toxicity | up to 3 years
  To evaluate early and late toxicity according to the NCI-CTC
Quality of Life evaluation (EORTC QLQ-C30 and QLQ-LC13) | up to 3 years
  To evaluate the quality of life at inclusion, at the end oh chemotherapy, 2 months after the radiotherapy and every 3 months until end of study